CLINICAL TRIAL: NCT01786772
Title: Neuromuscular Consequences of Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT12-16517
Record Dates: First submitted 2012-12-07; First posted 2013-02-08 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Tear of Fibrocartilage of Joint
Keywords: arthroscopic partial meniscectomy; meniscus; quadriceps strength; quadriceps voluntary activation; cryotherapy; compression; vasopneumatic compression; intermittent pneumatic compression
MeSH Terms: interventions — Cryotherapy; Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryotherapy and compression (Experimental): Cryotherapy and intermittent pneumatic compression will be applied to the knee joint using a recirculating compression unit and knee sleeve. This unit will recirculate water which is between 1-3° C. Circumferential intermittent pneumatic compression to the knee joint (5 to 50 mm Hg) will be applied in conjunction with cryotherapy. The duration of intervention will be 20 minutes.
  Interventions: Other: Cryotherapy and compression
- Cryotherapy (Active Comparator): Cryotherapy will be applied to the knee joint using a recirculating compression unit and knee sleeve. This unit will recirculate water which is between 1-3° C. The duration of intervention will be 20 minutes.
  Interventions: Other: Cryotherapy

INTERVENTIONS:
Other: Cryotherapy and compression — Cryotherapy and intermittent pneumatic compression will be applied to the knee joint using a recirculating compression unit and knee sleeve. This unit will recirculate water which is between 1-3° C. Circumferential intermittent pneumatic compression to the knee joint (5 to 50 mm Hg) will be applied in conjunction with cryotherapy. The duration of intervention will be 20 minutes.
  Other Names: Cryotherapy and intermittent pneumatic compression; Cryotherapy and vasopneumatic compression; Gameready
  Arms: Cryotherapy and compression
Other: Cryotherapy — Cryotherapy will be applied to the knee joint using a recirculating compression unit and knee sleeve. This unit will recirculate water which is between 1-3° C. The duration of intervention will be 20 minutes.
  Other Names: Ice; Gameready
  Arms: Cryotherapy

SUMMARY:
To determine changes in quadriceps muscle function following the application of ice and compression to the knee.

DETAILED DESCRIPTION:
Novel rehabilitation methods, that specifically target decreased muscle activation due to joint pathology prior to strength training, have elicited greater improvements in muscle function and self-reported disability compared to traditional therapies. Preliminary evidence suggests applying cryotherapy to a joint prior to exercise can increase quadriceps activation. It is unknown if applying cryotherapy and intermittent pneumatic compression can also increase quadriceps force output and voluntary activation. The purpose of this study is to determine changes in quadriceps force output and voluntary activation following the application of cryotherapy and compression. The investigators hypothesize there will be an increase in quadriceps force output and voluntary activation following the application of cryotherapy and compression.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-65 years
* BMI < 30
* Candidate for arthroscopic knee surgery to address meniscus pathology or arthroscopic knee surgery within the past 2 years.

Exclusion Criteria:

* Participants who are outside of age range
* Ligamentous insufficiency or repair
* Participants with traumatic spine or lower extremity injury within past 6 months
* Participants who have had previous adverse reactions to electrical stimulation or cryotherapy (i.e. burns, hypersensitivity)
* Medical conditions which would be contraindications to electrical stimulation or transcranial magnetic stimulation, including cardiac pacemaker, metal implants in the head, current pregnancy, neurological disorders, and history of seizures
* Participants who are unable to give consent or are unable to understand procedures of experiment.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in quadriceps force output and voluntary activation | Baseline and immediately following intervention (Single Study Visit)
  Quadriceps activation will be estimated by utilizing the burst-superimposition technique on a maximum voluntary isometric contraction (MVIC) and during a resting condition. The burst-superimposition technique provides the muscle with a percutaneous stimulus to recruit any remaining muscle fibers which have not been stimulated.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Grindstaff, PhD, PT, ATC, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States